CLINICAL TRIAL: NCT01909713
Title: Tolerability of a Foaming Facial Cleanser and Moisturizer SPF 30 in a Pediatric Population (7-11) With Acne Prone Skin.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.SRE.04.US10245
Record Dates: First submitted 2013-07-01; First posted 2013-07-26 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2013-12

CONDITIONS: Acne Prone Skin
Keywords: acne, pediatric
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Facial Cleanser and Moisturizer SPF 30 (Experimental): All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days.
  Interventions: Drug: Facial Cleanser and Moisturizer SPF 30

INTERVENTIONS:
Drug: Facial Cleanser and Moisturizer SPF 30 — Cetaphil® DermaControl™ Foam Wash and Moisturizer SPF 30
  Other Names: Cetaphil® DermaControl™ skin care products

SUMMARY:
The purpose of this study is to determine the tolerability of Cetaphil® DermaControl™ Foam Wash and Moisturizer SPF 30 in pediatric subjects (7-11) with acne prone skin.

DETAILED DESCRIPTION:
This was a open-label, single center study conducted in the United States that evaluated the tolerability of Cetaphil® DermaControl™ skin care products used at least once daily for 22 days in male and female subjects age 7 to 11 with acne prone skin. There were 4 visits during the course of the study: screening (within 7 days of visit 1), visit 1(baseline /day1), visit 2 (day 8), and visit 3 (day 22/exit). Tolerability assessments were performed by a board certified dermatologist at all visits. Subjects completed the baseline skin care regimen questionnaire at visit 1. Hydration assessments were competed at visits 1, 2, and 3. A subject satisfaction questionnaire was completed at visit 3. Adverse event assessments were conducted for all subjects at every clinic visit after informed consent/assent was signed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 7-11 years of age
* Subjects with acne-prone skin [Global severity of acne (GSA) Score of 1 (almost clear) or 2 (mild) and any oiliness evaluation score or GSA Score of 0 (none) with an oiliness evaluation score greater than or equal to 1 (mild)]

Exclusion Criteria:

* Subjects with any visible skin condition or facial hair that could interfere with the evaluations
* Subjects taking other medications, supplements, or non-prescription treatments that, in the opinion of the principal investigator/board certified dermatologist, could interfere with the test results including any regimen of steroidal/non steroidal anti-inflammatory drugs or antihistamines
* Subjects currently under the treatment for asthma or diabetes (insulin-dependent only)
* Subjects with abnormal pigmented vascular skin lesions, abnormal skin pigmentation, or body art (tattoos, permanent or temporary) on the face, which could interfere with subsequent evaluations of dermal responsiveness

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren Winkelman, MD, MBA, PhD, Study Director — Galderma R&D
Locations (1):
- RCTS, Inc., Irving, Texas, United States

REFERENCES:
- [Derived] Hensley D, Meckfessel MH. Tolerability of a Skin Care Regimen Formulated for Acne-Prone Skin in Children. Pediatr Dermatol. 2015 Jul-Aug;32(4):501-5. doi: 10.1111/pde.12607. Epub 2015 May 14. PMID 25973678

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetaphil® DermaControl™ Regimen.: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days.
  Facial Cleanser and Moisturizer SPF 30: Cetaphil® DermaControl™ Foam Wash and Moisturizer SPF 30
Period: Overall Study
Arm/Group | Cetaphil® DermaControl™ Regimen.
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetaphil® DermaControl™ Regimen.
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (1.5)
Age, Customized [Median (Full Range); unit: years] | 9.0 [7.0 to 11.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 22
  More than one race | 2
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Normal Skin Type [Number; unit: participants] | 35
Fitzpatrick Skin Type [Number; unit: participants] — Fitzpatrick Skin Type Classification I Always burns; never tans II Burns easily; tans minimally III Burns moderately; tans gradually to light brown IV Burns minimally; tans well to moderate brown V Rarely burns; tans profusely to dark brown VI Never burns; tans profusely to black
  participants
    II | 7
    III | 5
    IV | 3
    V | 12
    VI | 8
Global Severity of Acne [Number; unit: participants]
  Clear | 1
  Almost Clear | 27
  MIld | 7
Oiliness Evaluation Score [Number; unit: participants]
  Not Oily | 28
  Mildly Oily | 7

OUTCOME MEASURES:

1. Primary Outcome: Cutaneous Tolerability Based on Visual Inspection - Erythema
Description: Cutaneous tolerability based on visual inspection (investigator reported severity scale) was assessed at visit 1 (day 1), visit 2 (day 8), and visit 3 (day 22). Erythema: 0 = none, no observable redness; 1 = very mild, slight redness, spotty or diffuse; 2 = mild, moderate redness; 3 = moderate, intense; 4 = severe, fiery red with edema.
Time Frame: Week 3
Measure: Number; unit: participants
Groups:
- Baseline: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days and were assessed for tolerability at baseline, week 1, and week 3. This arm shows the results from baseline.
- Week 1: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days and were assessed for tolerability at baseline, week 1, and week 3. This arm shows the results from week 1.
- Week 3: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days and were assessed for tolerability at baseline, week 1, and week 3. This arm shows the results from week 3.
- Worst Post Baseline: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days and were assessed for tolerability at baseline, week 1, and week 3. This arm shows the worst post baseline results for all time ponts collected.
Arm/Group | Baseline | Week 1 | Week 3 | Worst Post Baseline
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  None | 29 | 33 | 30 | 29
  Very Mild | 6 | 2 | 4 | 5
  Mild | 0 | 0 | 1 | 1

2. Secondary Outcome: Cutaneous Tolerability Based on Subject and Parent/Legally Authorized Representative Interview - Itching
Description: Cutaneous tolerability based on visual inspection (investigator reported severity scale) was assessed at visit 1 (day 1), visit 2 (day 8), and visit 3 (day 22). Itching: 0 = none, no itching; 1 = mild, slight itching, not really bothersome; 2 = moderate, definite itching that is somewhat bothersome; 3 = severe, intense itching that may interrupt daily activities and/or sleep
Time Frame: Week 3
Measure: Number; unit: participants
Arm/Group | Baseline | Week 1 | Week 3 | Worst Post Baseline
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  None | 33 | 31 | 34 | 30
  Mild | 2 | 4 | 1 | 5

3. Primary Outcome: Cutaneous Tolerability Based on Visual Inspection - Edema
Description: Cutaneous tolerability based on visual inspection (investigator reported severity scale) was assessed at visit 1 (day 1), visit 2 (day 8), and visit 3 (day 22). Edema: 0 = none; 1 = mild; 2 = moderate; 3 = intense.
Time Frame: Week 3
Measure: Number; unit: participants
Arm/Group | Baseline | Week 1 | Week 3 | Worst Post Baseline
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  None | 35 | 35 | 34 | 34
  Mild | 0 | 0 | 1 | 1

4. Primary Outcome: Cutaneous Tolerability Based on Visual Inspection - Dryness
Description: Cutaneous tolerability based on visual inspection (investigator reported severity scale) was assessed at visit 1 (day 1), visit 2 (day 8), and visit 3 (day 22). Dryness: 0 = no observable scaling; 1 = fine flakes/scaling; 2 = moderate flakes/scaling; 3 = larger flakes/severe scaling.
Time Frame: Week 3
Measure: Number; unit: participants
Arm/Group | Baseline | Week 1 | Week 3 | Worst Post Baseline
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  No Observable Scaling | 34 | 33 | 32 | 32
  Fine Flakes/Scaling | 1 | 2 | 3 | 3

5. Primary Outcome: Cutaneous Tolerability Based on Visual Inspection - Roughness
Description: Cutaneous tolerability based on visual inspection (investigator reported severity scale) was assessed at visit 1 (day 1), visit 2 (day 8), and visit 3 (day 22). Roughness: 1 - no roughness, skin is fine, silky smooth, 2 - firm (not too rough, not too smooth), 3 - coarse, rough skin, 4 - leathery, flaky skin.
Time Frame: Week 3
Measure: Number; unit: participants
Arm/Group | Baseline | Week 1 | Week 3 | Worst Post Baseline
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  No Roughness, Skin is Fine, Silky Smooth | 35 | 34 | 35 | 34
  Coarse, Rough Skin | 0 | 1 | 0 | 1

6. Secondary Outcome: Cutaneous Tolerability Based on Subject and Parent/Legally Authorized Representative Interview - Burning
Description: Cutaneous tolerability based on visual inspection (investigator reported severity scale) was assessed at visit 1 (day 1), visit 2 (day 8), and visit 3 (day 22). Burning: 0 = none, no burning; 1 = mild, slight burning sensation, not really bothersome; 2 = moderate, definite warm, burning sensation that is somewhat bothersome; 3 = severe, hot burning sensation that causes definite discomfort and may interrupt daily activities and/or sleep
Time Frame: Week 3
Measure: Number; unit: participants
Arm/Group | Baseline | Week 1 | Week 3 | Worst Post Baseline
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  None | 35 | 33 | 33 | 31
  Mild | 0 | 2 | 2 | 4

7. Secondary Outcome: Cutaneous Tolerability Based on Subject and Parent/Legally Authorized Representative Interview - Stinging
Description: Cutaneous tolerability based on visual inspection (investigator reported severity scale) was assessed at visit 1 (day 1), visit 2 (day 8), and visit 3 (day 22). Stinging: 0 = none, no stinging; 1 = mild, slight stinging sensation, not really bothersome; 2 = moderate, definite stinging sensation that is somewhat bothersome; 3 = severe, stinging sensation that causes definite discomfort and may interrupt daily activities and/or sleep
Time Frame: Week 3
Measure: Number; unit: participants
Arm/Group | Baseline | Week 1 | Week 3 | Worst Post Baseline
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  None | 35 | 34 | 35 | 34
  Mild | 0 | 1 | 0 | 1

8. Secondary Outcome: Cutaneous Tolerability Based on Subject and Parent/Legally Authorized Representative Interview - Tightness
Description: Cutaneous tolerability based on visual inspection (investigator reported severity scale) was assessed at visit 1 (day 1), visit 2 (day 8), and visit 3 (day 22). Tightness: 0 = none, no tightness; 1 = mild, slight tightness, not really bothersome; 2 = moderate, definite tightness sensation that is somewhat bothersome; 3 = severe, tightness sensation that causes definite discomfort and may interrupt daily activities and/or sleep
Time Frame: Week 3
Measure: Number; unit: participants
Arm/Group | Baseline | Week 1 | Week 3 | Worst Post Baseline
Number analyzed (Participants) | 35 | 35 | 35 | 35
participants
  None | 35 | 35 | 35 | 35
  Mild | 0 | 0 | 0 | 0

9. Secondary Outcome: Barrier Function (TEWL)
Description: Barrier function was assessed by measuring transepidermal water loss (TEWL) at visit 1 (day 1), visit 2 (day 8), and visit 3 (day 22). TEWL measures water loss through the epidermis (for example, by evaporation). Measuring TEWL is a well-established way to assess the skin's water-barrier function. High TEWL values indicate impaired skin barrier function; low values indicate normal barrier function.
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: g/m2/h
Groups:
- Baseline: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days. TEWL was assessed at baseline, week 1, and week 3. This arm shows the results from baseline.
- Week 1: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days, TEWL was assessed at baseline, week 1, and week 3. This arm shows the results from week 1.
- Week 3: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days. TEWL was assessed at baseline, week 1, and week 3. This arm shows the results from week 3.
Arm/Group | Baseline | Week 1 | Week 3
Number analyzed (Participants) | 35 | 35 | 35
g/m2/h | 8.89 (3.01) | 11.41 (5.22) | 11.29 (3.25)

10. Secondary Outcome: Hydration (Corneometry)
Description: Hydration was assessed using corneometry at visit 1 (day 1), visit 2 (day 8), and visit 3 (day 22). Corneometry measures the hydration status of the skin. An increase in corneometry values indicates an increase in the hydration status of the skin, and vice versa. The test is procedure specific, so results are reported in "arbitrary units."
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- Baseline: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days. Hydration as assessed using corneometry at baseline, week 1, and week 3. This arm shows the results from baseline.
- Week 1: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days. Hydration as assessed using corneometry at baseline, week 1, and week 3.This arm shows the results from week 1.
- Week 3: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days. Hydration as assessed using corneometry at baseline, week 1, and week 3. This arm shows the results from week 3.
Arm/Group | Baseline | Week 1 | Week 3
Number analyzed (Participants) | 35 | 35 | 35
arbitrary units | 55.75 (11.24) | 56.51 (12.00) | 48.28 (12.47)

11. Secondary Outcome: Subject Satisfaction Questionnaire - Face Wash
Description: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days. Patient satisfaction questions were asked for the face wash at study end (day 22).
Time Frame: Day 22
Measure: Number; unit: participants
Groups:
- I Liked Using the Face Wash; The Face Wash Was Easy to Use; The Face Wash Made my Skin Feel Clean; The Face Wash Rinsed Easily Off my Skin; I Would Keep Using the Face Wash: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days. Patient satisfaction questions were asked for the face wash at study end (day 22).
- I Liked the Face Wash Better Than What I Was Using Before: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days. Patient satisfaction questions were asked for the face wash at study end (day 22). Subjects were only required to respond to this question if they had used a face wash previously.
Arm/Group | I Liked Using the Face Wash | The Face Wash Was Easy to Use | The Face Wash Made my Skin Feel Clean | The Face Wash Rinsed Easily Off my Skin | I Would Keep Using the Face Wash | I Liked the Face Wash Better Than What I Was Using Before
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
participants
  Yes | 34 | 35 | 35 | 32 | 30 | 6
  No | 1 | 0 | 0 | 3 | 5 | 0
  Missing | 0 | 0 | 0 | 0 | 0 | 29

12. Secondary Outcome: Subject Satisfaction Questionnaire - Moisturizer
Description: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days. Patient satisfaction questions were asked for the moisturizer at study end (day 22).
Time Frame: Day 22
Measure: Number; unit: participants
Groups:
- I Liked Using the Lotion; The Lotion Smelled Good; The Lotion Spread Easily on my Skin; The Lotion Made my Skin Feel Soft; I Would Keep Using the Lotion: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days. Patient satisfaction questions were asked for the moisturizer at study end (day 22).
- I Liked the Lotion Better Than What I Was Using Before: All subjects used Cetaphil® DermaControl™ Oil Control Foam Wash and Cetaphil® DermaControl™ Oil Control Moisturizer SPF 30 at least once daily for 22 days. Patient satisfaction questions were asked for the moisturizer at study end (day 22). Subjects were only required to respond to this question if they had used a moisturizer previously.
Arm/Group | I Liked Using the Lotion | The Lotion Smelled Good | The Lotion Spread Easily on my Skin | The Lotion Made my Skin Feel Soft | I Would Keep Using the Lotion | I Liked the Lotion Better Than What I Was Using Before
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
participants
  Yes | 34 | 28 | 35 | 33 | 30 | 4
  No | 1 | 7 | 0 | 2 | 5 | 0
  Missing | 0 | 0 | 0 | 0 | 0 | 31

ADVERSE EVENTS:
Time Frame: There were 3 visits during the course of the study: visit 1(baseline/day1), visit 2 (day 8), and visit 3 (day 22/exit). Adverse event assessments were conducted for all subjects at every clinic visit after informed consent/assent was signed.
Arm/Group | Cetaphil® DermaControl™ Regimen.
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 11/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetaphil® DermaControl™ Regimen. (N=35)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Pityriasis alba (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Impetigo (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less